CLINICAL TRIAL: NCT03892447
Title: A 52-week Multicenter, Randomized, Double-blind, Prospective Study to Evaluate Comparative Effectiveness and Safety of Alprostadil Injection,Sodium Ferulate and Dopamine Injection in Pediatric Acute Kidney Injury
Brief Title: The Comparative Effectiveness of Alprostadil,Sodium Ferulate and Dopamine in Pediatric Acute Kidney Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yubin Wu, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJES001
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Children AKI Patients
Keywords: AKI; Child; Alprostadil; Sodium Ferulate; Dopamine
MeSH Terms: interventions — Alprostadil; ferulic acid; Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alprostadil (Experimental): Alprostadil 0.2~0.3ug/kg.h,iv,1h/d,14d; Dopamine3～5 ug/kg·min,iv,3 h/d,14d
  Interventions: Drug: Alprostadil; Drug: Dopamine
- Sodium Ferulate (Active Comparator): Sodium Ferulate 2~6mg/kg.d,iv,14d; Dopamine3～5 ug/kg·min,iv,3 h/d,14d
  Interventions: Drug: Sodium Ferulate; Drug: Dopamine

INTERVENTIONS:
Drug: Alprostadil — Alprostadil 0.2~0.3ug/kg.h,iv,1h/d,14d
  Arms: Alprostadil
Drug: Sodium Ferulate — Sodium Ferulate 2~6mg/kg.d,iv,14d
  Arms: Sodium Ferulate
Drug: Dopamine — Dopamine3～5 ug/kg·min,iv,3 h/d,14d

SUMMARY:
Acute kidney injury (AKI) is a pervasive clinical event in children.It has been independently associated with prolonged hospital stays, risk of in-hospital death and future progression to chronic kidney disease. Except for removal of nephrotoxic agents and optimization of supportive care,there are still no other effective therapeutic options recommended by recent guidelines. Renal ischemia is the main mechanism of AKI, the improving microcirculation therapy would be the effective management to improve the outcome of AKI in children.

Dopamine is a vasodilating drug that in small doses improves renal circulation. Alprostadil have been used in chronic arterial occlusion and Sodium Ferulate in ischemic cerebral vascular disease,they have a similar therapeutic effect of anti-platelet aggregation and vasodilation. Recent research shows that alprostadil might be associated with a significant reduction in postcontrast Scr, blood urine nitrogen (BUN) and Cystatin C (CysC) level and decrease the incidence of contrast-induced nephropathy.The investigators speculate that Alprostadil,Sodium Ferulate and dopamine would be effective in treating AKI in children.

This is a prospective, multicenter, randomized, double-blind, 52-week study. The purpose of this study is to evaluate the comparative effectiveness and safety of Alprostadil,Sodium Ferulate and dopamine in improving the outcome of AKI in children.

DETAILED DESCRIPTION:
This study aims to explore the effective treatment of pediatric AKI and improve the outcome. It is a 52-week multicenter, randomized, double-blind,prospective study to evaluate comparative effectiveness and safety of alprostadil injection,sodium ferulate and dopamine injection. This study plans to recruit 8 to 10 centers, with 300 participants randomly divided into 3 groups and given respectively Alprostadil 0.2~0.3ug/kg.h,iv,1h/d,14d,Sodium Ferulate2~6mg/kg.d,iv,14d,Dopamine3~5ug/kg .min,iv,3h/d,14d.Time of outcome measurement is 1w,2w,4w,24w,52w. Primary Outcome Measures is The change of Serum creatinin from baseline, estimated glomerular filtration rate (eGFR) and urine volume in the participants after the use of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent signed and dated by participants and/or their guardians
2. male or female, Asian.
3. Aged from 1 to 18 years.
4. Patients meet the AKI diagnosis criteria of 2012 Kidney Disease: Improving Global Outcome (SKDIGO) Guideline

Exclusion Criteria:

1. prerenal or postrenal failure
2. Patients need renal replacement therapy
3. Patients with hemorrhagic disorders
4. Patients in shock
5. Patients with multiple organ failure
6. History of Alprostadil or Sodium Ferulate or dopamine sensitivity
7. Patients with heart failure
8. Patients with peptic ulcer
9. Patients with glaucoma
10. Patients with interstitial pneumonia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum creatinin | baseline, 52 weeks
  The change of Serum creatinin from baseline after the use of the study drug.
eGFR | baseline, 52 weeks
  The change of eGFR from baseline after the use of the study drug. eGFR (ml/min/1.73m2)=K×L/SCr. L: Height(cm), SCr: serum creatinin (umol/L),K:36.5
Urine volume | baseline, 52 weeks
  The change of urine volume from baseline after the use of the study drug.

SECONDARY OUTCOMES:
Urinary markers：White Blood Cell (WBC) | baseline, 52 weeks
  Obtained through routine urine examination.
Urinary markers：Red Blood Cell (RBC) | baseline, 52 weeks
  Obtained through routine urine examination.
Urinary markers：Urine protein | baseline, 52 weeks
  Obtained through routine urine examination.
Serum urea | baseline, 52 weeks
  Obtained through renal function test.
Serum Cystatin | baseline, 52 weeks
  Obtained through renal function test.
Three dimensional(3D) color ultrasound Imaging | baseline, 52 weeks
  Size of kidneys,Blood flow of renal arteries.
Blood pressure | baseline, 52 weeks
Duration of hospital stays | baseline, 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shenjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
Dear Sir/Madam Our study receives a grant from China Ministry of Science and Technology. We cannot decide whether the data could be shared. Hope you can understand.

REFERENCES:
- See also: 2012 SKDIGO Guideline — http://kdigo.org/